CLINICAL TRIAL: NCT06184737
Title: iSIPsmarter: A Pilot RCT to Evaluate a Technology-based Behavioral Intervention to Reduce Sugary Beverages Among Black Adults
Brief Title: iSIPsmarter: A Pilot RCT to Evaluate a Web-based Behavioral Intervention to Reduce Sugary Beverages Among Black Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of North Carolina (Other)
Responsible Party: Principal Investigator, Jamie Zoellner, PhD RD, Director, Community Based Health Equity Program, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22130
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Diet Habit; Sugar-Sweetened Beverages
Keywords: sugar-sweetened beverages; weight; health disparities; self-monitoring; internet intervention; e/m health; text messaging
MeSH Terms: conditions — Feeding Behavior; Body Weight | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iSIPsmarter (Experimental): iSIPsmarter is a technology-based behavioral and health literacy intervention. It is comprised of six Internet-delivered Cores, an integrated short message service (SMS) strategy to engage users in tracking SSB behaviors, and the incorporation of a cellular enabled scale for in-home weight tracking. Participants will be prompted (via email or text) to self-monitor their sugar-sweetened beverage intake. iSIPsmarter is a highly interactive, structured, and self-guided program that uses strategies previously proven to promote behavior change. iSIPsmarter also incorporates a stepped care approach to re-engage users who struggle to complete components.
  Interventions: Behavioral: iSIPsmarter
- Patient Education (PE) (Active Comparator): The PE website will include scientifically accurate information that is typical of nutrition education websites and will include information about SSB recommendations, types of SSB and portion size, SSB-related health risks, energy balance information, identifying personal motivators and barriers to reducing SSB intake, interpreting SSB nutrition labels, and recognizing media influences and misclaims in SSB advertisements, as well as printable forms to track SSB and weight. Unlike iSIPsmarter, the content will not be tailored and will be presented all at once.
  Interventions: Behavioral: Patient Education (PE)

INTERVENTIONS:
Behavioral: iSIPsmarter — iSIPsmarter is a technology-based behavioral and health literacy intervention. It is comprised of six Internet-delivered Cores, an integrated short message service (SMS) strategy to engage users in tracking SSB behaviors, and the incorporation of a cellular enabled scale for in-home weight tracking. Participants will be prompted (via email or text) to self-monitor their sugar-sweetened beverage intake. iSIPsmarter is a highly interactive, structured, and self-guided program that uses strategies previously proven to promote behavior change. iSIPsmarter also incorporates a stepped care approach to re-engage users who struggle to complete components.
  Arms: iSIPsmarter
Behavioral: Patient Education (PE) — The PE website will include scientifically accurate information that is typical of nutrition education websites and will include information about SSB recommendations, types of SSB and portion size, SSB-related health risks, energy balance information, identifying personal motivators and barriers to reducing SSB intake, interpreting SSB nutrition labels, and recognizing media influences and misclaims in SSB advertisements, as well as printable forms to track SSB and weight. Unlike iSIPsmarter, the content will not be tailored and will be presented all at once.
  Arms: Patient Education (PE)

SUMMARY:
The proposed pilot randomized controlled trial (RCT) will enroll 24 Black adults. The overall goal is to examine the preliminary efficacy of iSIPsmarter in a 2 group [iSIPsmarter vs. static Patient Education (PE) website] by 4 assessment (Pre, 3-, 6- and 18-month follow-up) design. The generated pilot data will allow us to better understand efficacy and engagement outcomes among Black participants. We anticipate trends that iSIPsmarter will be more efficacious at reducing SSB consumption than a PE website at post assessment.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults, identify as Black, > or equal to 18 years of age, consume >200 kcals of SSB/day, ability and willingness to access an internet-enabled device at least one time per week and receive SMS-based reminder prompts

Exclusion Criteria:

* non-English speaking adults, do not identify as Black, <18 years of age, consume <200 kcals of SSB/day, inability and willingness to access an internet-enabled device at least one time per week and receive SMS-based reminder prompts. Also, only one person per household is eligible to participate in the trial

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline sugar-sweetened beverage at 9-weeks | Baseline, 9-weeks (immediate-post follow-up)
  Measured using the Beverage Questionnaire 15 (BEVQ-15)

SECONDARY OUTCOMES:
Change from baseline dietary quality as measured by the components of the Healthy Eating Index (HEI) at 9-weeks, 6-months and 18 months | Baseline, 9-weeks (immediate-post follow-up), 6-months, 18 months
  2 unannounced recalls (one weekend and one weekday) using state-of-the-art Nutrition Data System for Research (NDSR) software and multiple pass methods. HEI indicators will be extracted from the NDSR system and examined for changes in the total HEI score, on a 100-point continuous scale (higher scores reflective higher diet quality).
Change from baseline weight at 9-weeks, 6-months and 18 months | Baseline, 9-weeks (immediate-post follow-up), 6-months, 18 months
  Cellular enabled in-home ©BodyTrace digital scale
Change from baseline overall quality of life at 9-weeks, 6-months and 18 months | Baseline, 9-weeks (immediate-post follow-up), 6-months, 18 months
  Using the Center's for Disease (CDC) Healthy Days Core Module
Change from baseline sugar-sweetened beverage at 6-months and 18 months | Baseline, 6-months, 18 months
  Measured using the BEVQ-15

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Zoellner, PhD, Principal Investigator — University of Virginia; Lee Ritterband, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No